CLINICAL TRIAL: NCT03039023
Title: Effects of Choline From Eggs vs. Supplements on the Generation of TMAO in Humans (EGGS)
Brief Title: Effects of Choline From Eggs vs. Supplements on the Generation of TMAO in Humans
Acronym: EGGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Staff, Cardiovascular Medicine, The Cleveland Clinic; Staff, Cellular and Molecular Medicine, The Cleveland Clinic Lerner Research Institute, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1048
Record Dates: First submitted 2017-01-19; First posted 2017-02-01 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Risk Factor
Keywords: TMAO; choline; eggs; gastrointestinal microbiome; healthy volunteers
MeSH Terms: interventions — Choline; Phosphatidylcholines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Whole Hardboiled Eggs (Experimental): Subjects will consume four (4) pre-cooked, pre-peeled whole hardboiled eggs per day for 28 days.
  Interventions: Other: Pre-cooked, pre-peeled whole hardboiled eggs
- Choline Bitartrate Tablets (Experimental): Subjects will consume two (2) 500mg choline bitartrate tablets per day for 28 days.
  Interventions: Dietary Supplement: Choline Bitartrate
- Hardboiled Eggs + Choline Bitartrate Tablets (Experimental): Subjects will consume both four (4) whole, pre-cooked, pre-peeled hardboiled eggs and two (2) 500mg choline bitartrate tablets per day for 28 days.
  Interventions: Dietary Supplement: Choline Bitartrate; Other: Pre-cooked, pre-peeled whole hardboiled eggs
- Egg Whites + Choline Bitartrate Tablets (Experimental): Subjects will consume both the egg whites (no yolks) of four (4) pre-cooked, pre-peeled hardboiled eggs and two (2) 500mg choline bitartrate tablets per day for 28 days.
  Interventions: Dietary Supplement: Choline Bitartrate; Other: Egg whites from pre-cooked, pre-peeled hardboiled eggs
- Phosphatidylcholine Capsules (Experimental): Subjects will consume six (6) 420 mg phosphatidylcholine capsules by mouth per day for 28 days.
  Interventions: Dietary Supplement: Phosphatidylcholine capsules

INTERVENTIONS:
Dietary Supplement: Choline Bitartrate — 500mg choline bitartrate tablets
  Arms: Choline Bitartrate Tablets; Egg Whites + Choline Bitartrate Tablets; Hardboiled Eggs + Choline Bitartrate Tablets
Other: Pre-cooked, pre-peeled whole hardboiled eggs — Obtained from a commercial source.
  Arms: Hardboiled Eggs + Choline Bitartrate Tablets; Whole Hardboiled Eggs
Other: Egg whites from pre-cooked, pre-peeled hardboiled eggs — Egg whites from pre-cooked, pre-peeled hardboiled eggs. The yolks are removed and discarded.
  Arms: Egg Whites + Choline Bitartrate Tablets
Dietary Supplement: Phosphatidylcholine capsules — 420 mg phosphatidylcholine capsules obtained from a commercial source.
  Arms: Phosphatidylcholine Capsules

SUMMARY:
The investigators are interested in learning more about choline, a nutrient required by the body. The body does make some choline, but it does not make enough to support health and the rest must be acquired through diet. Eggs, and especially egg yolks, are a major dietary source of choline. Choline can also be given as a dietary supplement. Ingestion of choline supplements has been linked to an increased concentration of a compound called TMAO (trimethylamine N-oxide). Elevated TMAO levels have been linked to higher heart disease risk. With this study, the investigators hope to learn whether there is a difference in the way your body responds to the ingestion of a choline supplement versus the choline found within eggs.

DETAILED DESCRIPTION:
The principal goal for the study is to examine whether there is a difference between the ingestion of choline through supplements versus choline found within eggs on plasma TMAO levels. The investigators have previously shown that dietary intake of trimethylamines, including the choline group of phosphatidylcholine (PC), is mechanistically linked to cardiovascular disease risk and that the metabolism of these trimethylamine nutrients in humans is modulated by the intestinal microbes (gut microbes). Additionally, extensive animal studies link an essential role of gut microbiota to the metabolism of choline and the production of metabolites that promote / accelerate atherosclerotic processes. The investigators have also recently shown a 10-fold increase in plasma TMAO levels following supplementation with choline bitartrate supplements. However, another pilot study by a collaborator (unpublished) did not show the same increase in plasma TMAO levels following the ingestion of whole eggs, a major dietary source of choline. Therefore, with this study the investigators wish to examine the differences, if any, between the ingestion of an equivalent mass of total choline in the free form (as bitartrate salt) as a supplement vs. within whole eggs.

Eggs, and specifically the egg yolk, contain a large amount of total choline. However, egg white contains potential anti-microbial peptides that could influence gut microbial composition and function, and therefore impact conversion of choline into TMA and TMAO observed in subjects. Therefore, the investigators hypothesize that the consumption of whole eggs (hardboiled) will not elevate plasma TMAO levels to the same extent as a comparable amount of total choline ingested in capsule form as the choline bitartrate salt. The investigators further hypothesize that the consumption of egg white with choline bitartrate tablets may result in less of a rise in TMAO levels than ingestion of the choline bitartrate supplement alone.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or above.
* Willing to remain on aspirin or stay off aspirin or aspirin products for 1 week prior to starting the study and throughout the study period.
* Able to provide informed consent and comply with study protocol.
* Able to be off all other supplements during the study period.

Exclusion Criteria:

* Significant chronic illness.
* Active infection or received antibiotics within 1 month of study enrollment.
* Use of over-the-counter probiotic within the past month
* Chronic gastrointestinal disorders, such as ulcerative colitis or Crohn's disease.
* Allergy to eggs or lactose.
* Having undergone bariatric procedures or surgeries such as gastric banding or bypass.
* Pregnancy.
* Any condition that, in the judgment of the Investigator, would place a patient at undue risk by being enrolled in the trial or cause inability to comply with the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Rebouche CJ, Chenard CA. Metabolic fate of dietary carnitine in human adults: identification and quantification of urinary and fecal metabolites. J Nutr. 1991 Apr;121(4):539-46. doi: 10.1093/jn/121.4.539. PMID 2007906
- [Background] Bidulescu A, Chambless LE, Siega-Riz AM, Zeisel SH, Heiss G. Repeatability and measurement error in the assessment of choline and betaine dietary intake: the Atherosclerosis Risk in Communities (ARIC) study. Nutr J. 2009 Feb 20;8:14. doi: 10.1186/1475-2891-8-14. PMID 19232103
- [Derived] Wilcox J, Skye SM, Graham B, Zabell A, Li XS, Li L, Shelkay S, Fu X, Neale S, O'Laughlin C, Peterson K, Hazen SL, Tang WHW. Dietary Choline Supplements, but Not Eggs, Raise Fasting TMAO Levels in Participants with Normal Renal Function: A Randomized Clinical Trial. Am J Med. 2021 Sep;134(9):1160-1169.e3. doi: 10.1016/j.amjmed.2021.03.016. Epub 2021 Apr 17. PMID 33872583
- See also: Patterson K, Bhagwat S, Williams J, Howe J, and Holden J. USDA Database for the Choline Content of Common Foods, Release Two. January 2008. — https://data.nal.usda.gov/system/files/Choln02.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Started | 19 | 20 | 17 | 20 | 10
Completed | 18 | 20 | 16 | 18 | 10
Not Completed | 1 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules | Total
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10 | 82
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25.5 [23.3 to 28.8] | 27.0 [23.0 to 37.0] | 37.0 [24.0 to 50.3] | 30.0 [25.0 to 35.8] | 31.5 [25.8 to 47.3] | 28.0 [24.0 to 38.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 15 | 10 | 6 | 48
  Male | 10 | 11 | 1 | 8 | 4 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 0 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 2 | 1 | 7
  White | 13 | 15 | 16 | 16 | 7 | 67
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 20 | 16 | 18 | 10 | 82
TMAO at Baseline [Median (Inter-Quartile Range); unit: uM] | 2.0 [1.4 to 3.5] | 1.9 [1.4 to 3.4] | 2.3 [1.5 to 2.8] | 2.6 [1.8 to 5.3] | 2.8 [2.0 to 5.1] | 2.3 [1.5 to 3.5]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Plasma Levels of Fasting Trimethylamine-N-oxide (TMAO), a Choline Metabolite
Description: Changes in levels of non-labeled TMAO from baseline to end-of-study (day 28) as measured by established techniques by mass spectrometry.
Time Frame: Baseline, 28 days
Population: All participants with TMAO measured at baseline and Day 28.
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
uM
  Baseline | 2.0 [1.4 to 3.5] | 1.9 [1.4 to 3.4] | 2.3 [1.5 to 2.8] | 2.6 [1.8 to 5.3] | 2.8 [2.0 to 5.1]
  Day 28 | 2.3 [1.9 to 3.7] | 11.1 [7.1 to 25.4] | 12.3 [5.1 to 26.5] | 28.1 [9.2 to 44.1] | 3.4 [2.6 to 7.1]
Statistical Analysis 1: Comparison: Whole Hardboiled Eggs; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.20, Wilcoxon signed-rank test — A p-value <0.05 was considered significant
Statistical Analysis 2: Comparison: Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 3: Comparison: Hardboiled Eggs + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 4: Comparison: Egg Whites + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 5: Comparison: Phosphatidylcholine Capsules; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.27, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant

2. Primary Outcome: Changes in Platelet Function With Increased Choline Intake
Description: The activation and functioning of platelets within a single subject will be compared before and after increased choline intake.
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: aggregation percentage
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 10
aggregation percentage
  Baseline | 2.6 [1.4 to 5.3] | 2.6 [1.2 to 7.2] | 2.3 [1.6 to 3.0] | 3.0 [2.3 to 5.0] | 2.8 [2.0 to 4.0]
  Day 28 | 3.6 [2.5 to 7.7] | 12.8 [7.6 to 27.2] | 12.3 [6.1 to 25.7] | 29.4 [17.9 to 43.3] | 3.4 [2.6 to 7.1]
Statistical Analysis 1: Comparison: Whole Hardboiled Eggs; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.10, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 2: Comparison: Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.0002, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 3: Comparison: Hardboiled Eggs + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.01, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 4: Comparison: Egg Whites + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.006, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 5: Comparison: Phosphatidylcholine Capsules; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.79, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant

3. Secondary Outcome: Changes in Levels of Fasting Trimethylamine-N-oxide (TMAO) in 24-hour Urine Collections
Description: Changes in levels of non-labeled TMAO from baseline to Day 28 measured by established mass spectrometry techniques.
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: mg in 24 hours
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 19 | 16 | 18 | 10
mg in 24 hours
  Baseline | 24.3 [13.0 to 44.3] | 26.2 [15.6 to 40.3] | 27.5 [9.1 to 36.2] | 29.3 [18.4 to 45.9] | 15.8 [12.9 to 35.6]
  Day 28 | 28.5 [23.1 to 36.7] | 139.0 [90.1 to 308.9] | 221.8 [166.3 to 294.3] | 186.9 [91.2 to 232.4] | 33.1 [19.9 to 64.6]
Statistical Analysis 1: Comparison: Whole Hardboiled Eggs; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.28, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 2: Comparison: Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 3: Comparison: Hardboiled Eggs + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 4: Comparison: Egg Whites + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 5: Comparison: Phosphatidylcholine Capsules; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.11, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant

4. Secondary Outcome: Changes in Plasma Levels of Fasting Choline
Description: Fasting plasma levels of choline from samples obtained at baseline and at day 28 were compared.
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
uM
  Baseline | 8.3 [6.6 to 10.2] | 7.5 [6.5 to 9.3] | 8.5 [7.6 to 11.2] | 9.5 [7.6 to 11.6] | 7.6 [6.7 to 9.1]
  Day 28 | 10.9 [8.9 to 12.4] | 12.9 [10.8 to 16.0] | 14.0 [11.7 to 15.7] | 12.8 [10.2 to 14.1] | 10.6 [9.2 to 11.6]
Statistical Analysis 1: Comparison: Whole Hardboiled Eggs; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.005, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 2: Comparison: Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 3: Comparison: Hardboiled Eggs + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 4: Comparison: Egg Whites + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.009, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 5: Comparison: Phosphatidylcholine Capsules; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.04, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant

5. Secondary Outcome: Changes in Plasma Levels of Fasting Carnitine.
Description: Fasting plasma levels of carnitine from samples obtained at baseline and at day 28 were compared.
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
uM
  Baseline | 19.1 [16.3 to 22.8] | 21.2 [16.6 to 25.1] | 21.5 [16.8 to 24.8] | 21.1 [16.5 to 26.6] | 23.4 [17.8 to 28.1]
  Day 28 | 19.4 [13.4 to 27.9] | 18.7 [15.5 to 21.0] | 15.6 [10.9 to 19.4] | 18.9 [15.2 to 23.2] | 20.8 [19.1 to 27.5]
Statistical Analysis 1: Comparison: Whole Hardboiled Eggs; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.93, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 2: Comparison: Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.01, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 3: Comparison: Hardboiled Eggs + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.003, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 4: Comparison: Egg Whites + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.04, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 5: Comparison: Phosphatidylcholine Capsules; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.99, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant

6. Secondary Outcome: Changes in Plasma Levels of Fasting Betaine.
Description: Fasting plasma levels of betaine from samples obtained at baseline and at day 28 were compared.
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
uM
  Baseline | 28.1 [23.6 to 48.3] | 38.2 [28.7 to 48.7] | 30.7 [18.4 to 35.7] | 38.7 [23.3 to 47.7] | 33.6 [23.3 to 45.0]
  Day 28 | 39.7 [29.4 to 55.5] | 69.0 [54.4 to 82.2] | 46.9 [33.9 to 67.5] | 59.8 [41.6 to 65.6] | 46.3 [28.3 to 64.0]
Statistical Analysis 1: Comparison: Whole Hardboiled Eggs; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.02, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 2: Comparison: Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 3: Comparison: Hardboiled Eggs + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p < 0.0001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 4: Comparison: Egg Whites + Choline Bitartrate Tablets; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.001, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant
Statistical Analysis 5: Comparison: Phosphatidylcholine Capsules; Test type: Equivalence — For equivalence testing, the difference was assumed to be 0; p = 0.02, Wilcoxon Signed Rank test — A p-value <0.05 was considered significant

7. Secondary Outcome: Changes in Lipid Profile, Total Cholesterol
Description: Changes in total cholesterol levels between baseline and Day 28
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
mg/dL
  Baseline | 156 [145 to 175] | 180 [147 to 201] | 187 [172 to 204] | 186 [150 to 189] | 175 [159 to 217]
  Day 28 | 158 [136 to 180] | 172 [157 to 191] | 198 [168 to 221] | 178 [157 to 193] | 172 [151 to 213]

8. Secondary Outcome: Changes in Lipid Profile, HDL
Description: Changes in measured HDL levels between baseline and Day 28
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
mg/dL
  Baseline | 48 [44 to 66] | 49 [40 to 60] | 57 [50 to 65] | 48 [39 to 63] | 61 [49 to 65]
  Day 28 | 49 [44 to 65] | 51 [44 to 60] | 56 [49 to 74] | 50 [41 to 57] | 62 [42 to 64]

9. Secondary Outcome: Changes in Lipid Profile, LDL
Description: Changes in measured LDL levels between baseline and Day 28
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
mg/dL
  Baseline | 91 [72 to 102] | 90 [80 to 124] | 108 [98 to 120] | 104 [86 to 124] | 107 [90 to 137]
  Day 28 | 86 [71 to 110] | 94 [82 to 119] | 118 [87 to 132] | 101 [87 to 121] | 106 [79 to 136]

10. Secondary Outcome: Changes in Lipid Profile, Triglycerides
Description: Changes in measured triglyceride levels between baseline and Day 28
Time Frame: Baseline, Day 28
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
Number analyzed (Participants) | 18 | 20 | 16 | 18 | 10
mg/dL
  Baseline | 86 [70 to 112] | 106 [74 to 134] | 103 [89 to 125] | 122 [52 to 156] | 74 [67 to 89]
  Day 28 | 100 [57 to 116] | 96 [82 to 141] | 97 [80 to 111] | 109 [69 to 170] | 84 [67 to 96]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during study participation, up to 30 days from enrollment.
Arm/Group | Whole Hardboiled Eggs | Choline Bitartrate Tablets | Hardboiled Eggs + Choline Bitartrate Tablets | Egg Whites + Choline Bitartrate Tablets | Phosphatidylcholine Capsules
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/17 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/17 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/17 | 0/20 | 0/10

LIMITATIONS AND CAVEATS:
Small sample sizes within each group created uneven distributions of some baseline characteristics; participants' dietary intake beyond the assigned interventions was not controlled during the study period; using only healthy controls makes the translatability of the results to other patient populations, like those with impaired renal function, unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT03039023/Prot_SAP_000.pdf